CLINICAL TRIAL: NCT00324129
Title: A Phase I Study of MGCD0103 Given as a Three-Times Weekly Oral Dose In Patients With Leukemia Or Myelodysplastic Syndromes
Brief Title: A Phase I Study of MGCD0103 Given Three-Times Weekly In Patients With Leukemia Or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Gregory Reid, Chief Medical Officer, MethylGene, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-003
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: Leukemia; Myelodysplastic Syndromes; Phase I
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MGCD0103

INTERVENTIONS:
Drug: MGCD0103 — MGCD0103 given orally three times per week.

SUMMARY:
In this study, MGCD0103, a new anticancer drug under investigation, is given three times weekly to patients with leukemia or myelodysplastic syndromes.

DETAILED DESCRIPTION:
Phase I dose escalating study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of one of the following:

  * relapsed or refractory AML or ALL that has failed to respond to standard therapy, has progressed despite standard therapy
  * relapsed or refractory Myelodysplastic Syndromes
  * previously untreated AML or Myelodysplastic Syndromes in patients > 60 years of age who refused or are not candidates for induction chemotherapy
* Patients with relapsed or refractory CML that has failed to respond to Imatinib therapy or standard therapy, has progressed despite standard therapy, or for which no standard therapy exists
* ECOG performance status of 0, 1, or 2
* Age ≥ 18 years
* Patients or their legal representative must be able to read, understand, and sign a written informed consent (approved by the IRB/EC) prior to study entry

Exclusion Criteria:

* Patients with a history of another cancer other than basal cell carcinoma or cervical intraepithelial neoplasia
* Pregnant or lactating women
* Patients and their partners, if either are of childbearing potential, not using adequate birth control measures throughout the study and for 90 days following the last dose of study medication
* Patients with known meningeal metastasis(es)
* Patients with active or uncontrolled infections, or with a fever >38.5 C
* Patients with serious illnesses, medical conditions, or other medical history, which would be likely to interfere with a patient's participation in the study
* Patients who have been treated with any investigational drug or anti-cancer therapy within 30 days of study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-02; Primary Completion 2006-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 1 year (anticipated)
Pharmacokinetics | 1 year (anticipated)

SECONDARY OUTCOMES:
Clinical Response | 1 year (anticipated)
Dose limiting toxicities | 1 year (anticipated)
Pharmacodynamics (histone acetylation, biomarkers) | 1 year (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (3):
- Anderson Cancer Center, Houston, Texas, United States
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Sir Mortimer Davis-Jewish General Hospital, Montreal, Quebec